CLINICAL TRIAL: NCT04507360
Title: Enhancing Engagement With Digital Mental Health Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Mental Health America (Other); Talkspace (Industry); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Tim Althoff, Assistant Professor, Computer Science and Engineering, University of Washington
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Health Services Research
Other Study IDs: STUDY00010958; 1R01MH125179-01 (NIH)
Record Dates: First submitted 2020-08-05; First posted 2020-08-11 (Actual); Results first posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Engagement, Patient
Keywords: Digital Mental Health
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Intervention Model Description: The investigators will conduct focus groups applying user-centered design strategies to identify and co-build potentially effective engagement strategies for particular client subtypes. The investigators anticipate enrolling 10,000 Mental Health America consumers in Study 1 (the sequential multiple assignment randomized trial; SMART), with a subset of 250 participating in Study 2, a randomized controlled trial of an Artificial Intelligence (AI)-assisted self-help tool compared to a non-AI self help tool and to psychoeducational materials only control group.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Study 1, Demographic Survey + Generic Response + Generic Resources (Experimental): This arm included participants who completed the Demographics Survey (stage 1 randomization).
  The Generic Response + Generic Resources condition (stage 2 randomization) will feature the response-as-usual on Mental Health America (MHA)'s website and the four generic resource pages on MHA's website.
  Interventions: Behavioral: Study 1, Demographics Survey; Behavioral: Study 1, Generic Response; Behavioral: Study 1, Generic Resources
- Study 1, Demographic Survey + Generic Response + Tailored Resources by Demographics (Experimental): This arm included participants who completed the Demographics Survey (stage 1 randomization).
  The Generic Response + Tailored Resources by Demographics condition (stage 2 randomization) will feature the response-as-usual on Mental Health America (MHA)'s website and resources tailored to two demographics. People who endorse being Lesbian, Gay, Bisexual, Transgender, or Queer (LGBTQ) will receive 4 resources associated with LGBTQ issues. People who endorse being 8-17, 18-24, 25-44, or 45+ years of age will receive 4 resources used by people in those age groups. If someone enters both age and LGBTQ status, they will be provided with 2 resources tailored to age and 2 resources tailored to LGBTQ status, randomly chosen.
  Interventions: Behavioral: Study 1, Demographics Survey; Behavioral: Study 1, Generic Response; Behavioral: Study 1, Tailored Resources by Demographics
- Study 1, Next Steps Survey + Generic Response + Generic Resources (Experimental): This arm included participants who completed the Next Steps Survey (stage 1 randomization).
  The Generic Response + Generic Resources condition (stage 2 randomization) will feature the response-as-usual on Mental Health America (MHA)'s website and the four generic resource pages on MHA's website.
  Interventions: Behavioral: Study 1, Next Steps Survey; Behavioral: Study 1, Generic Response; Behavioral: Study 1, Generic Resources
- Study 1, Next Steps Survey + Generic Response + Tailored Resources by Desired Resources (Experimental): This arm included participants who completed the Next Steps Survey (stage 1 randomization).
  The Generic Response + Tailored Resources by Desired Resources condition (stage 2 randomization) will feature the response-as-usual on Mental Health America (MHA)'s website and 4 resources tailored to a survey question that asks participants what they would like to do next on the website after screening is complete (e.g., "Learn more about depression", "Take another mental health test")
  Interventions: Behavioral: Study 1, Next Steps Survey; Behavioral: Study 1, Generic Response; Behavioral: Study 1, Tailored Resources by Desired Resources
- Study 1, Next Steps Survey + Tailored Response + Generic Resources (Experimental): This arm included participants who completed the Next Steps Survey (stage 1 randomization).
  The Tailored Response + Generic Resources condition (stage 2 randomization) will feature a response tailored to screening status (above or below criteria for depression) and expressed need for mental health support (e.g., "We're so glad to hear you're open to exploring how to improve your mental health. People who score with minimum or mild depression often notice that symptoms can get worse in the weeks after taking a Depression test.") They will also receive the 4 generic resources.
  Interventions: Behavioral: Study 1, Next Steps Survey; Behavioral: Study 1, Generic Resources; Behavioral: Study 1, Tailored Response
- Study 1, Next Steps Survey + Tailored Response + Tailored Resources by Desired Resources (Experimental): This arm included participants who completed the Next Steps Survey (stage 1 randomization).
  The Tailored Response + Tailored Resources by Desired Resources condition (stage 2 randomization) will feature a response tailored to screening status (above or below criteria for depression) and expressed need for mental health support, and will receive resources tailored to a survey question that asks participants what they would like to do next on the website after screening is complete (e.g., "Learn more about depression", "Take another mental health test").
  Interventions: Behavioral: Study 1, Next Steps Survey; Behavioral: Study 1, Tailored Response; Behavioral: Study 1, Tailored Resources by Desired Resources
- Study 2, Control (Experimental): Participants in the Do-It-Yourself (DIY) control group will receive psychoeducation materials in week 0. They will view content as usual (no DIY) and will receive surveys from week 1 to week 4 and follow-up surveys in week 5 and at the end of week 8.
  Interventions: Behavioral: Study 2, Control
- Study 2, DIY tool without AI (Experimental): Participants in the Do-It-Yourself (DIY) tool without Artificial Intelligence (AI) group will be instructed to use the DIY tool 3 times a week. They will receive surveys from week 1 to week 4 and follow-up surveys in week 5 and at the end of week 8.
  Interventions: Behavioral: Study 2, DIY tool without AI
- Study 2, DIY tool with AI (Experimental): Participants in the Do-It-Yourself (DIY) tool with Artificial Intelligence (AI) group will be instructed to use the DIY tool with AI 3 times a week. They will receive surveys from week 1 to week 4 and follow-up surveys in week 5 and at the end of week 8.
  Interventions: Behavioral: Study 2, DIY tool with AI
- Study 1, Demographic Survey (Experimental): This arm included participants who were randomized to the Demographics Survey (stage 1 randomization) and were not randomized to a stage 2 condition (i.e., did not view screening results page on which stage 2 randomization occurred).
  Interventions: Behavioral: Study 1, Demographics Survey
- Study 1, Next Steps Survey (Experimental): This arm included participants who were randomized to the Next Steps Survey (stage 1 randomization) and were not randomized to a stage 2 condition (i.e., did not view screening results page on which stage 2 randomization occurred).
  Interventions: Behavioral: Study 1, Next Steps Survey

INTERVENTIONS:
Behavioral: Study 1, Demographics Survey — Participants will be shown a demographics survey (e.g., age range, gender, income).
  Arms: Study 1, Demographic Survey; Study 1, Demographic Survey + Generic Response + Generic Resources; Study 1, Demographic Survey + Generic Response + Tailored Resources by Demographics
Behavioral: Study 1, Next Steps Survey — Participants will be shown the Next Steps Survey, which includes 2 items assessing intended next steps on the Mental Health America (MHA) website (e.g., take another mental health test, find a treatment provider near you) and perceived need (yes, no, or I don't know) in addition to the Demographics Survey items.
  Arms: Study 1, Next Steps Survey; Study 1, Next Steps Survey + Generic Response + Generic Resources; Study 1, Next Steps Survey + Generic Response + Tailored Resources by Desired Resources; Study 1, Next Steps Survey + Tailored Response + Generic Resources; Study 1, Next Steps Survey + Tailored Response + Tailored Resources by Desired Resources
Behavioral: Study 1, Generic Response — Participants will be provided with the generic/current response to screening.
  Arms: Study 1, Demographic Survey + Generic Response + Generic Resources; Study 1, Demographic Survey + Generic Response + Tailored Resources by Demographics; Study 1, Next Steps Survey + Generic Response + Generic Resources; Study 1, Next Steps Survey + Generic Response + Tailored Resources by Desired Resources
Behavioral: Study 1, Generic Resources — Participants will be provided with links to a list of 4 generic Mental Health America (MHA) resources.
  Arms: Study 1, Demographic Survey + Generic Response + Generic Resources; Study 1, Next Steps Survey + Generic Response + Generic Resources; Study 1, Next Steps Survey + Tailored Response + Generic Resources
Behavioral: Study 1, Tailored Response — Participants will be provided with a response to screening that is tailored to the match between screening score (above or below depression criteria) and expressed need for mental health support (yes, no, or I don't know).
  Arms: Study 1, Next Steps Survey + Tailored Response + Generic Resources; Study 1, Next Steps Survey + Tailored Response + Tailored Resources by Desired Resources
Behavioral: Study 1, Tailored Resources by Demographics — Participants will be provided with links to Mental Health America (MHA) resources tailored to sexuality (Lesbian, Gay, Bisexual, Transgender, or Queer) status and age range.
  Arms: Study 1, Demographic Survey + Generic Response + Tailored Resources by Demographics
Behavioral: Study 1, Tailored Resources by Desired Resources — Participants will be provided with links to Mental Health America (MHA) resources aligned with their expressed interest (e.g., additional screening, self help tools).
  Arms: Study 1, Next Steps Survey + Generic Response + Tailored Resources by Desired Resources; Study 1, Next Steps Survey + Tailored Response + Tailored Resources by Desired Resources
Behavioral: Study 2, Control — Participants in the Do-It-Yourself (DIY) control group will receive psychoeducation materials in W0. They will view content as usual (no DIY).
  Arms: Study 2, Control
Behavioral: Study 2, DIY tool without AI — Participants in the Do-It-Yourself (DIY) tool without Artificial Intelligence (AI) group will be instructed to use the DIY tool 3 times a week.
  Arms: Study 2, DIY tool without AI
Behavioral: Study 2, DIY tool with AI — Participants in the Do-It-Yourself (DIY) tool with Artificial Intelligence (AI) group will be instructed to use the DIY tool with AI 3 times a week.
  Arms: Study 2, DIY tool with AI

SUMMARY:
This proposal is a partnership between Mental Health America (MHA), a nonprofit mental health advocacy and resource organization, Talkspace (TS), a for-profit, online digital psychotherapy organization, and the University of Washington's Schools of Medicine and Computer Science Engineering (UW). The purpose of this partnership is to create a digital mental health research platform leveraging MHA and TS's marketing platforms and consumer base to describe the characteristics of optimal engagement with digital mental health treatment, and to identify effective, personalized methods to enhance motivation to engage in digital mental health treatment in order to improve mental health outcomes. These aims will be met by identifying and following at least 100,000 MHA and TS consumers over the next 4 years, apply machine learning approaches to characterizing client engagement subtypes, and apply micro-randomized trials to study the effectiveness of motivational enhancement strategies and response to digital mental health treatment.

DETAILED DESCRIPTION:
Digital mental health (DMH) is the use of technology to improve population well-being through rapid disease detection, outcome measurement, and care. Although several randomized clinical trials have demonstrated that digital mental health tools are highly effective, most consumers do not sustain their use of these tools. The field currently lacks an understanding of DMH tool engagement, how engagement is associated with well-being, and what practices are effective at sustaining engagement. In this partnership between Mental Health America (MHA), Talkspace (TS), and the University of Washington (UW), the investigators propose a naturalistic and experimental, theory-driven program of research, with the aim of understanding 1) how consumer engagement in self-help and clinician assisted DMH varies and what engagement patterns exist, 2) the association between patterns of engagement and important consumer outcomes, and 3) the effectiveness of personalized strategies for optimal engagement with DMH treatment.

This study will prospectively follow a large, naturalistic sample of MHA and TS consumers, and will apply machine learning, user-centered design strategies, and micro randomized and sequential multiple assignment randomized trials (SMART) to address these aims. As is usual practice for both platforms, consumers will complete online mental health screening and assessment, and the investigators will be able to classify participants by disease status and symptom severity. The sample that the investigators will be working with will not be limited by diagnosis or co-morbidities. Participants will enter the MHA and TS platforms prospectively over 4 years. For aim 1, participant data will be analyzed statistically to reveal differences in engagement and dropout across groups based on demographics, symptoms and platform activity. For aim 2, the investigators will use supervised machine learning techniques to identify subtypes based on consumer demographics, engagement patterns with DMH, reasons for disengagement, success of existing MHA and TS engagement strategies, and satisfaction with the DMH tools, that are predictive of future engagement patterns. Finally, based on the outcomes from aim 2, in aim 3a the investigators will conduct focus groups applying user centered design strategies to identify and co-build potentially effective engagement strategies for particular client subtypes. The investigators will then conduct a series of micro-randomized and SMART trials to determine which theory-driven engagement strategies, co-designed with users, have the greatest fit with subtypes developed under aim 2. The investigators will test the effectiveness of these strategies to 1) prevent disengagement from those who are more likely to have poor outcomes after disengagement, 2) improve movement from motivation to volition and, 3) enhance optimal dose of DMH engagement and consequently improve mental health outcomes. These data will be analyzed using longitudinal mixed effects models with effect coding to estimate the effectiveness of each strategy on client engagement behavior and mental health outcomes.

The purpose of aim 3b is to identify effective engagement strategies tailored to client needs and demographics to increase MHA website engagement, and to better understand how self-help mental health resources can help people overcome negative thinking and support healthier thought processes. The investigators will compare effective engagement strategies tailored to subtypes developed under aim 2 to study the mediated impact of engagement strategies on consumer mental health outcomes. The study team will determine if engagement strategies targeted to consumer engagement subtype will enhance engagement and in turn result in improved clinical outcomes. These will be compared to generic strategies that are not subtype targeted.

All aim 3b activities will occur with MHA, broken down into two parts: (Study 1) a sequential multiple assignment randomized trial (SMART) and (Study 2) a Do-It-Yourself (DIY) tool longitudinal randomized control trial (RCT). Study 1 will use a SMART to examine methods to optimize engagement with MHA's website, and Study 2 will recruit participants for a longitudinal month-long study where they are randomly assigned to a control group, the use of a DIY tool without Artificial Intelligence (AI), or the use of a DIY tool with AI to examine the efficacy of using a digital tool to improve mental health functioning. An AI tool that uses machine learning/Natural Language Processing (NLP)/AI methods was developed to personalize and tailor an intervention to improve engagement and completion outcomes. The study focuses on a specific, popular DIY tool that teaches cognitive restructuring. Pilot work showed that (1) engagement and completion rates on DIY tools can be low, and (2) a pilot AI tool had significantly higher engagement and completion rates. These differences may arise due to AI support, User Interface/User Experience/design differences, other factors, or a combination thereof. Additionally, the efficacy of the digital tool to improve mental health functioning is unknown. Study 2 will recruit participants who will be randomly assigned to one of three groups for a longitudinal month-long study: thrice-weekly DIY tool use with AI, without AI, or a control group.

ELIGIBILITY:
Inclusion Criteria:

* Phase 3b Study 1 (Sequential Multiple Assignment Randomized Trial; SMART): Users of the Mental Health America (MHA) website, engaging from Internet Protocol (IP) addresses in the United States, who have chosen to start the PHQ-9 depression screener in English. Must be those who can read English.
* Phase 3b Study 2 (Do-It-Yourself; DIY): Patient Health Questionnaire (PHQ)-9 or Generalized Anxiety Disorder (GAD)-7 score of 10 or greater, users of MHA website, 18 years of age or older.

Exclusion Criteria:

* Phase 3b Study 1 (SMART): None
* Phase 3b Study 2 (DIY): Younger than 18 years old, Non-English or Non-Spanish speaking, PHQ-9 less than 10, outside of US, have more than a little familiarity with the concept of cognitive reframing.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 78390 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pullmann, PhD, Principal Investigator — University of Washington
Locations (3):
- United States (3):
  - Groop Internet Platform DBA Talkspace, New York, New York
  - Mental Health America, Alexandria, Virginia
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Zech JM, Johnson M, Pullmann MD, Hull TD, Althoff T, Munson SA, Fridling N, Litvin B, Wu J, Arean PA. An Integrative Engagement Model of Digital Psychotherapy: Exploratory Focus Group Findings. JMIR Form Res. 2023 Apr 26;7:e41428. doi: 10.2196/41428. PMID 37099363

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Time points are not applicable to Study 1. Study 1: stage 1 conditions include 1) Demographics Survey and 2) Next Steps Survey; stage 2 conditions include 1) Generic Response + Generic Resources, 2) Generic Response + Tailored Resources by Demographics, 3) Generic Response + Tailored Resources by Desired Resources, 4) Tailored Response + Generic Resources, and 5) Tailored Response + Tailored Resources by Desired Resources.
Pre-assignment Details: Study 2:
  Started: participants we reached out to for filling out weekly survey or using Do-It-Yourself (DIY) tool.
  Completed: participants who completed weekly survey or finished using DIY tool at least once.
  Not Completed: participants who did not complete weekly survey and did not finish using DIY tool even once.
  Completion was not required to continue participation in the study; number "Started" at each time is always the same as the total number of participants enrolled in the study.
Groups:
- Study 2, Control: Participants in the Do-It-Yourself (DIY) control group will receive psychoeducation materials in W0. They will view content as usual (no DIY) and will receive surveys from W1 to W4 and follow-up surveys in W5 and at the end of W8.
  Study 2, Control: Participants in the Do-It-Yourself (DIY) control group will receive psychoeducation materials in W0. They will view content as usual (no DIY).
- Study 2, DIY Tool Without AI: Participants in the Do-It-Yourself (DIY) tool without Artificial Intelligence (AI) group will be instructed to use the DIY tool 3 times a week. They will receive surveys from W1 to W4 and follow-up surveys in W5 and at the end of W8.
  Study 2, DIY tool without AI: Participants in the Do-It-Yourself (DIY) tool without Artificial Intelligence (AI) group will be instructed to use the DIY tool 3 times a week.
- Study 2, DIY Tool With AI: Participants in the Do-It-Yourself (DIY) tool with Artificial Intelligence (AI) group will be instructed to use the DIY tool with AI 3 times a week. They will receive surveys from W1 to W4 and follow-up surveys in W5 and at the end of W8.
  Study 2, DIY tool with AI: Participants in the Do-It-Yourself (DIY) tool with Artificial Intelligence (AI) group will be instructed to use the DIY tool with AI 3 times a week.
Period: Baseline
Arm/Group | Study 1, Demographic Survey | Study 1, Next Steps Survey | Study 1, Demographic Survey + Generic Response + Generic Resources | Study 1, Demographic Survey + Generic Response + Tailored Resources by Demographics | Study 1, Next Steps Survey + Generic Response + Generic Resources | Study 1, Next Steps Survey + Generic Response + Tailored Resources by Desired Resources | Study 1, Next Steps Survey + Tailored Response + Generic Resources | Study 1, Next Steps Survey + Tailored Response + Tailored Resources by Desired Resources | Study 2, Control | Study 2, DIY Tool Without AI | Study 2, DIY Tool With AI
Started | 2490 | 2367 | 19250 | 19240 | 8743 | 8636 | 8454 | 8371 | 269 | 272 | 298
Completed | 2490 | 2367 | 19250 | 19240 | 8743 | 8636 | 8454 | 8371 | 269 | 272 | 298
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Week 1
Arm/Group | Study 1, Demographic Survey | Study 1, Next Steps Survey | Study 1, Demographic Survey + Generic Response + Generic Resources | Study 1, Demographic Survey + Generic Response + Tailored Resources by Demographics | Study 1, Next Steps Survey + Generic Response + Generic Resources | Study 1, Next Steps Survey + Generic Response + Tailored Resources by Desired Resources | Study 1, Next Steps Survey + Tailored Response + Generic Resources | Study 1, Next Steps Survey + Tailored Response + Tailored Resources by Desired Resources | Study 2, Control | Study 2, DIY Tool Without AI | Study 2, DIY Tool With AI
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 269 | 272 | 298
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 197 | 250 | 288
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 72 | 22 | 10
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 72 | 22 | 10
Period: Week 2
Arm/Group | Study 1, Demographic Survey | Study 1, Next Steps Survey | Study 1, Demographic Survey + Generic Response + Generic Resources | Study 1, Demographic Survey + Generic Response + Tailored Resources by Demographics | Study 1, Next Steps Survey + Generic Response + Generic Resources | Study 1, Next Steps Survey + Generic Response + Tailored Resources by Desired Resources | Study 1, Next Steps Survey + Tailored Response + Generic Resources | Study 1, Next Steps Survey + Tailored Response + Tailored Resources by Desired Resources | Study 2, Control | Study 2, DIY Tool Without AI | Study 2, DIY Tool With AI
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 269 | 272 | 298
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 148 | 187 | 216
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 121 | 85 | 82
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 121 | 85 | 82
Period: Week 3
Arm/Group | Study 1, Demographic Survey | Study 1, Next Steps Survey | Study 1, Demographic Survey + Generic Response + Generic Resources | Study 1, Demographic Survey + Generic Response + Tailored Resources by Demographics | Study 1, Next Steps Survey + Generic Response + Generic Resources | Study 1, Next Steps Survey + Generic Response + Tailored Resources by Desired Resources | Study 1, Next Steps Survey + Tailored Response + Generic Resources | Study 1, Next Steps Survey + Tailored Response + Tailored Resources by Desired Resources | Study 2, Control | Study 2, DIY Tool Without AI | Study 2, DIY Tool With AI
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 269 | 272 | 298
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 146 | 180 | 214
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 123 | 92 | 84
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 123 | 92 | 84
Period: Week 4
Arm/Group | Study 1, Demographic Survey | Study 1, Next Steps Survey | Study 1, Demographic Survey + Generic Response + Generic Resources | Study 1, Demographic Survey + Generic Response + Tailored Resources by Demographics | Study 1, Next Steps Survey + Generic Response + Generic Resources | Study 1, Next Steps Survey + Generic Response + Tailored Resources by Desired Resources | Study 1, Next Steps Survey + Tailored Response + Generic Resources | Study 1, Next Steps Survey + Tailored Response + Tailored Resources by Desired Resources | Study 2, Control | Study 2, DIY Tool Without AI | Study 2, DIY Tool With AI
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 269 | 272 | 298
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 138 | 157 | 196
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 131 | 115 | 102
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 131 | 115 | 102
Period: Week 5
Arm/Group | Study 1, Demographic Survey | Study 1, Next Steps Survey | Study 1, Demographic Survey + Generic Response + Generic Resources | Study 1, Demographic Survey + Generic Response + Tailored Resources by Demographics | Study 1, Next Steps Survey + Generic Response + Generic Resources | Study 1, Next Steps Survey + Generic Response + Tailored Resources by Desired Resources | Study 1, Next Steps Survey + Tailored Response + Generic Resources | Study 1, Next Steps Survey + Tailored Response + Tailored Resources by Desired Resources | Study 2, Control | Study 2, DIY Tool Without AI | Study 2, DIY Tool With AI
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 269 | 272 | 298
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 166 | 137 | 155
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 103 | 135 | 143
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 103 | 135 | 143
Period: Week 8
Arm/Group | Study 1, Demographic Survey | Study 1, Next Steps Survey | Study 1, Demographic Survey + Generic Response + Generic Resources | Study 1, Demographic Survey + Generic Response + Tailored Resources by Demographics | Study 1, Next Steps Survey + Generic Response + Generic Resources | Study 1, Next Steps Survey + Generic Response + Tailored Resources by Desired Resources | Study 1, Next Steps Survey + Tailored Response + Generic Resources | Study 1, Next Steps Survey + Tailored Response + Tailored Resources by Desired Resources | Study 2, Control | Study 2, DIY Tool Without AI | Study 2, DIY Tool With AI
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 269 | 272 | 298
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 130 | 127 | 146
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 139 | 145 | 152
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 139 | 145 | 152

BASELINE CHARACTERISTICS:
Groups:
- : Study 1, Next Steps Survey: This arm included participants who were randomized to the Next Steps Survey (stage 1 randomization) and were not randomized to a stage 2 condition (i.e., did not view screening results page on which stage 2 randomization occurred).
- Total: Total of all reporting groups
Arm/Group | Study 1, Demographic Survey | : Study 1, Next Steps Survey | Study 1, Demographic Survey + Generic Response + Generic Resources | Study 1, Demographic Survey + Generic Response + Tailored Resources by Demographics | Study 1, Next Steps Survey + Generic Response + Generic Resources | Study 1, Next Steps Survey + Generic Response + Tailored Resources by Desired Resources | Study 1, Next Steps Survey + Tailored Response + Generic Resources | Study 1, Next Steps Survey + Tailored Response + Tailored Resources by Desired Resources | Study 2, Control | Study 2, DIY Tool Without AI | Study 2, DIY Tool With AI | Total
Number analyzed (Participants) | 2490 | 2367 | 19250 | 19240 | 8743 | 8636 | 8454 | 8371 | 269 | 272 | 298 | 78390
Age, Customized [Count of Participants; unit: Participants]
  Under 18 years old | 1280 | 1147 | 8127 | 8385 | 3683 | 3695 | 3627 | 3581 | 0 | 0 | 0 | 33525
  18-24 years old | 518 | 517 | 4149 | 4047 | 1911 | 1902 | 1753 | 1842 | 50 | 47 | 51 | 16787
  25-44 years old | 428 | 457 | 4501 | 4411 | 2065 | 1950 | 2041 | 1968 | 137 | 153 | 173 | 18284
  45 years old and older | 207 | 187 | 2176 | 2101 | 931 | 942 | 900 | 841 | 82 | 72 | 74 | 8513
  Unknown or Not Reported | 57 | 59 | 297 | 296 | 153 | 147 | 133 | 139 | 0 | 0 | 0 | 1281
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 1450 | 1377 | 11558 | 11507 | 5233 | 5274 | 4973 | 4972 | 146 | 135 | 133 | 46758
  Male | 919 | 870 | 6979 | 6991 | 3131 | 3023 | 3113 | 3049 | 33 | 22 | 27 | 28157
  Nonbinary | 97 | 96 | 536 | 580 | 271 | 250 | 262 | 261 | 5 | 4 | 8 | 2370
  Unknown or not reported | 24 | 24 | 177 | 162 | 108 | 89 | 106 | 89 | 85 | 111 | 130 | 1105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 366 | 359 | 2590 | 2734 | 1264 | 1237 | 1184 | 1209 | 22 | 19 | 25 | 11009
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 158 | 139 | 137 | 434
  Unknown or Not Reported | 2124 | 2008 | 16660 | 16506 | 7479 | 7399 | 7270 | 7162 | 89 | 114 | 136 | 66947
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 75 | 59 | 392 | 397 | 181 | 196 | 175 | 196 | 2 | 1 | 5 | 1679
  Race: Asian | 267 | 237 | 1777 | 1755 | 821 | 777 | 784 | 733 | 12 | 10 | 3 | 7176
  Race: Native Hawaiian or Other Pacific Islander | 15 | 15 | 73 | 112 | 43 | 53 | 40 | 37 | 1 | 2 | 0 | 391
  Race: Black or African American | 190 | 250 | 1719 | 1683 | 766 | 825 | 767 | 772 | 11 | 5 | 9 | 6997
  Race: White | 1155 | 1040 | 10027 | 9977 | 4436 | 4344 | 4326 | 4201 | 142 | 138 | 135 | 39921
  Race: Middle Eastern or North African | 31 | 23 | 200 | 182 | 91 | 82 | 95 | 86 | 3 | 0 | 0 | 793
  Race: More than one race | 165 | 146 | 991 | 975 | 437 | 454 | 411 | 446 | 0 | 0 | 0 | 4025
  Race: Unknown or Not Reported | 128 | 138 | 872 | 791 | 423 | 401 | 397 | 425 | 98 | 116 | 146 | 3935
  Race: Other | 98 | 100 | 609 | 634 | 281 | 267 | 275 | 266 | 0 | 0 | 0 | 2530
  Race: Hispanic or Latino | 366 | 359 | 2590 | 2734 | 1264 | 1237 | 1184 | 1209 | 0 | 0 | 0 | 10943
Patient Health Questionnaire-9 [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire-9 (PHQ-9) consists of 9 depression items. Each item is associated with a Diagnostic and Statistical Manual (DSM) symptom of depression. Participants rate whether or not they have experienced the symptom over the last two weeks, with severity ratings of 0 to 3. Total scores range from 0 to 27, with higher scores indicating greater severity of depression symptoms. It is one of the few measures that is brief (it takes less than one minute to give) and has been found to have excellent sensitivity to change over time. Population: Study 1 and Study 2 baseline Patient Health Questionnaire-9 (PHQ-9) scores are presented separately in different rows.
  units on a scale
    Study 1: number analyzed (Participants) | 2490 | 2367 | 19250 | 19240 | 8743 | 8636 | 8454 | 8371 | 0 | 0 | 0 | 77551
    Study 1 | 16.02 (6.36) | 15.83 (6.38) | 15.83 (6.08) | 15.79 (6.09) | 15.90 (6.07) | 15.93 (6.11) | 15.85 (6.07) | 15.98 (6.10) |  |  |  | 15.86 (6.11)
    Study 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 269 | 272 | 298 | 839
    Study 2 |  |  |  |  |  |  |  |  | 17.69 (4.66) | 17.66 (4.86) | 17.97 (4.68) | 17.78 (4.73)
Generalized Anxiety Disorder-7 [Mean (Standard Deviation); unit: units on a scale] — The Generalized Anxiety Disorder-7 (GAD-7) is a 7- item screener for generalized anxiety. It consists of items related to Generalized Anxiety Disorder (GAD). Participants rate how much anxiety they have experienced in the last two weeks on a scale of 0 to 3. Total scores range from 0 to 21, with higher scores indicating greater severity of anxiety symptoms. The scale is a valid screener for GAD. Population: Data were not collected for Study 1. For Study 2, "Number Analyzed" includes participants who contributed data at baseline.
  units on a scale
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 268 | 271 | 298 | 837
    (all) |  |  |  |  |  |  |  |  | 14.29 (4.62) | 14.56 (4.14) | 14.38 (4.65) | 14.41 (4.48)

OUTCOME MEASURES:

1. Primary Outcome: Study 1: Mental Health America Disengagement (After Stage 1 Randomization)
Description: Proportion of users disengaging (i.e., by leaving the website; in contrast to clicking to view the screening results page or clicking another Mental Health America [MHA] link) after stage 1 randomization.
Time Frame: Through active web session, an average of 10 minutes
Population: Study 1 participants by stage 1 condition. Arms/Groups are combined by Demographics Survey and Next Steps survey because this outcome examined disengagement prior to stage 2 randomization.
Measure: Count of Participants; unit: Participants
Groups:
- Study 1, Demographics Survey (Stage 1 Randomization): This arm included participants who were randomized to receive the Demographics Survey after completing a screening tool on the Mental Health America (MHA) website. It includes 1) Study 1, Demographic Survey, 2) Study 1, Demographic Survey + Generic Response + Generic Resources, and 3) Demographic Survey + Generic Response + Tailored Resources by Demographics.
- Study 1, Next Steps Survey (Stage 1 Randomization): This arm included participants who were randomized to receive the Next Steps Survey after completing a screening tool on the Mental Health America (MHA) website. It includes 1) Study 1, Next Steps Survey, 2) Study 1, Next Steps Survey + Generic Response + Generic Resources, 3) Study 1, Next Steps Survey + Generic Response + Tailored Resources by Desired Resources, 4) Study 1, Next Steps Survey + Tailored Response + Generic Resources, and 5) Study 1, Next Steps Survey + Tailored Response + Tailored Resources by Desired Resources.
Arm/Group | Study 1, Demographics Survey (Stage 1 Randomization) | Study 1, Next Steps Survey (Stage 1 Randomization)
Number analyzed (Participants) | 40980 | 36571
Participants | 574 | 566

2. Primary Outcome: Study 1: Mental Health America Engagement, Clicks on Featured Resources (After Stage 2 Randomization)
Description: Proportion of users clicking featured resources (i.e., links to webpages on Mental Health America, featured below screening results) from the screening results page.
Time Frame: Through active web session, an average of 10 minutes
Population: Participants randomized to a stage 2 condition
Measure: Count of Participants; unit: Participants
Groups:
- Experimental: Study 1, Demographic Survey + Generic Response + Generic Resources: This arm included participants who completed the Demographics Survey (stage 1 randomization).
  The Generic Response + Generic Resources condition (stage 2 randomization) will feature the response-as-usual on Mental Health America (MHA)'s website and the four generic resource pages on MHA's website.
- Experimental: Study 1, Next Steps Survey + Generic Response + Generic Resources: This arm included participants who completed the Next Steps Survey (stage 1 randomization).
  The Generic Response + Generic Resources condition (stage 2 randomization) will feature the response-as-usual on Mental Health America (MHA)'s website and the four generic resource pages on MHA's website.
Arm/Group | Experimental: Study 1, Demographic Survey + Generic Response + Generic Resources | Study 1, Demographic Survey + Generic Response + Tailored Resources by Demographics | Experimental: Study 1, Next Steps Survey + Generic Response + Generic Resources | Study 1, Next Steps Survey + Generic Response + Tailored Resources by Desired Resources | Study 1, Next Steps Survey + Tailored Response + Generic Resources | Study 1, Next Steps Survey + Tailored Response + Tailored Resources by Desired Resources
Number analyzed (Participants) | 19250 | 19240 | 8743 | 8636 | 8454 | 8371
Participants | 2839 | 4517 | 1272 | 1457 | 1181 | 1507

3. Primary Outcome: Study 1: Mental Health America Engagement, Number of Webpages Clicked (After Stage 2 Randomization)
Description: Number of webpages clicked (including links to either featured and non-featured resources) after stage 2 randomization.
Time Frame: Through active web session, an average of 10 minutes
Population: Participants randomized to a stage 2 condition.
Measure: Mean (Standard Deviation); unit: Number of webpages
Arm/Group | Study 1, Demographic Survey + Generic Response + Generic Resources | Study 1, Demographic Survey + Generic Response + Tailored Resources by Demographics | Study 1, Next Steps Survey + Generic Response + Generic Resources | Study 1, Next Steps Survey + Generic Response + Tailored Resources by Desired Resources | Study 1, Next Steps Survey + Tailored Response + Generic Resources | Study 1, Next Steps Survey + Tailored Response + Tailored Resources by Desired Resources
Number analyzed (Participants) | 19250 | 19240 | 8743 | 8636 | 8454 | 8371
Number of webpages | 4.32 (12.86) | 5.05 (15.17) | 4.31 (11.66) | 4.43 (12.69) | 4.39 (13.07) | 4.12 (11.68)

4. Primary Outcome: Study 1: Mental Health America Disengagement (After Stage 2 Randomization)
Description: Proportion of users disengaging (i.e., by leaving the website; in contrast to clicking a link to a Mental Health America [MHA] webpage) after stage 2 randomization.
Time Frame: Through active web session, an average of 10 minutes
Population: Participants randomized to a stage 2 condition.
Measure: Count of Participants; unit: Participants
Arm/Group | Study 1, Demographic Survey + Generic Response + Generic Resources | Study 1, Demographic Survey + Generic Response + Tailored Resources by Demographics | Study 1, Next Steps Survey + Generic Response + Generic Resources | Study 1, Next Steps Survey + Generic Response + Tailored Resources by Desired Resources | Study 1, Next Steps Survey + Tailored Response + Generic Resources | Study 1, Next Steps Survey + Tailored Response + Tailored Resources by Desired Resources
Number analyzed (Participants) | 19250 | 19240 | 8743 | 8636 | 8454 | 8371
Participants | 9019 | 8532 | 4107 | 4100 | 3908 | 3891

5. Primary Outcome: Study 1: DIY Completion Rate (After Stage 2 Randomization)
Description: Number of participants who completed the Do-It-Yourself (DIY) tool.
Time Frame: Through active web session, an average of 10 minutes
Population: Participants randomized to a stage 2 condition who also accessed the Do-It-Yourself (DIY) tool by clicking on a content page.
Measure: Count of Participants; unit: Participants
Arm/Group | Study 1, Demographic Survey + Generic Response + Generic Resources | Study 1, Demographic Survey + Generic Response + Tailored Resources by Demographics | Study 1, Next Steps Survey + Generic Response + Generic Resources | Study 1, Next Steps Survey + Generic Response + Tailored Resources by Desired Resources | Study 1, Next Steps Survey + Tailored Response + Generic Resources | Study 1, Next Steps Survey + Tailored Response + Tailored Resources by Desired Resources
Number analyzed (Participants) | 3172 | 4204 | 1468 | 1489 | 1360 | 1445
Participants | 131 | 173 | 55 | 54 | 63 | 69

6. Primary Outcome: Study 2: Engagement (Dosage)
Description: Number of times using the Do-It-Yourself (DIY) tool
Time Frame: Week 1, Week 2, Week 3, Week 4
Population: "Overall Number of Participants Analyzed" includes participants who provided data (by finishing using the Do-It-Yourself [DIY] tool at least once) at any time point. "Number analyzed" includes participants who contributed data (finished used the DIY tool at least once) at that time point.
Measure: Mean (Standard Deviation); unit: usages
Arm/Group | Study 2, DIY Tool Without AI | Study 2, DIY Tool With AI
Number analyzed (Participants) | 223 | 249
usages
  Week 1: number analyzed (Participants) | 215 | 236
  Week 1 | 2.72 (1.48) | 2.99 (1.69)
  Week 2: number analyzed (Participants) | 157 | 179
  Week 2 | 1.98 (1.62) | 2.14 (1.68)
  Week 3: number analyzed (Participants) | 145 | 176
  Week 3 | 1.77 (1.65) | 2.14 (1.67)
  Week 4: number analyzed (Participants) | 125 | 157
  Week 4 | 1.63 (1.67) | 1.79 (1.63)
  Overall | 2.03 (1.66) | 2.26 (1.72)
Statistical Analysis 1: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference in "Overall" row; Test type: Superiority; Mean Difference (Final Values) = .23

7. Primary Outcome: Study 2: Tool Use Helpfulness
Description: Tool Use Helpfulness is measured using one item (Using the tool has been helpful to me in dealing with my negative thoughts and emotions) on a scale of 0 (strongly disagree) to 3 (strongly agree). Higher scores indicate better outcomes (helpfulness of the tool). Scores will be assessed using mean item-level scores. Note: includes 5 qualitative questions, not included here.
Time Frame: Week 1, Week 2, Week 3, Week 4
Population: "Overall Number of Participants Analyzed" includes participants who provided data at any time point. "Number analyzed" includes participants who contributed data at that time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study 2, DIY Tool Without AI | Study 2, DIY Tool With AI
Number analyzed (Participants) | 178 | 202
units on a scale
  Week 1: number analyzed (Participants) | 159 | 173
  Week 1 | 2.00 (0.75) | 1.99 (0.69)
  Week 2: number analyzed (Participants) | 117 | 124
  Week 2 | 1.88 (0.78) | 1.95 (0.74)
  Week 3: number analyzed (Participants) | 120 | 149
  Week 3 | 1.85 (0.83) | 1.83 (0.81)
  Week 4: number analyzed (Participants) | 113 | 132
  Week 4 | 1.82 (0.78) | 1.85 (0.83)

8. Primary Outcome: Study 2: Emotion Mechanisms
Description: Emotion mechanisms are measured using a 7-item scale. Each item is scored from 1 to 7. Total scores range from 7 to 49. Higher scores indicate better emotion mechanisms. Participants are asked about their emotions (e.g., hopefulness, worry, confidence, motivation) about their ability to address negative thoughts. Scores will be assessed using mean item-level and total scores.
  Item 1: How hopeful do you feel about the future? Item 2: How hopeful do you feel about managing negative thoughts? Item 3: How worried do you feel about managing negative thoughts? (reverse-coded) Item 4: How motivated are you to keep working on managing negative thinking? Item 5: How confident are you in your ability to identify thinking traps? Item 6: How confident are you in your ability to reframe negative thoughts? Item 7: How likely are you to recommend it to a friend?
Time Frame: Week 1, Week 2, Week 3, Week 4, Week 8
Population: "Overall Number of Participants Analyzed" includes participants who provided data at any time point. "Number analyzed" includes participants who contributed data at that time point. For "Total" score rows, "Number analyzed" includes participants who contributed sufficient item-level data to compute a total score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study 2, Control | Study 2, DIY Tool Without AI | Study 2, DIY Tool With AI
Number analyzed (Participants) | 219 | 196 | 219
units on a scale
  Week 1, Item 1: number analyzed (Participants) | 195 | 172 | 182
  Week 1, Item 1 | 3.66 (1.28) | 3.87 (1.43) | 3.77 (1.23)
  Week 1, Item 2: number analyzed (Participants) | 196 | 171 | 182
  Week 1, Item 2 | 3.62 (1.31) | 3.94 (1.31) | 3.85 (1.30)
  Week 1, Item 3: number analyzed (Participants) | 196 | 171 | 182
  Week 1, Item 3 | 3.56 (1.46) | 3.53 (1.42) | 3.51 (1.49)
  Week 1, Item 4: number analyzed (Participants) | 196 | 171 | 182
  Week 1, Item 4 | 5.32 (1.48) | 5.48 (1.43) | 5.19 (1.52)
  Week 1, Item 5: number analyzed (Participants) | 196 | 171 | 182
  Week 1, Item 5 | 4.19 (1.35) | 4.30 (1.47) | 4.12 (1.41)
  Week 1, Item 6: number analyzed (Participants) | 196 | 171 | 182
  Week 1, Item 6 | 3.66 (1.28) | 3.98 (1.53) | 3.90 (1.33)
  Week 1, Item 7: number analyzed (Participants) | 196 | 171 | 182
  Week 1, Item 7 | 4.80 (1.72) | 5.11 (1.62) | 4.85 (1.67)
  Week 1, Total: number analyzed (Participants) | 195 | 171 | 181
  Week 1, Total | 28.81 (6.13) | 30.18 (6.82) | 29.22 (6.24)
  Week 2, Item 1: number analyzed (Participants) | 145 | 118 | 126
  Week 2, Item 1 | 3.73 (1.37) | 4.03 (1.53) | 3.84 (1.36)
  Week 2, Item 2: number analyzed (Participants) | 145 | 118 | 126
  Week 2, Item 2 | 3.79 (1.31) | 4.14 (1.46) | 4.06 (1.26)
  Week 2, Item 3: number analyzed (Participants) | 145 | 118 | 126
  Week 2, Item 3 | 3.98 (1.51) | 3.86 (1.55) | 3.93 (1.33)
  Week 2, Item 4: number analyzed (Participants) | 145 | 118 | 126
  Week 2, Item 4 | 5.14 (1.53) | 5.42 (1.36) | 5.43 (1.39)
  Week 2, Item 5: number analyzed (Participants) | 145 | 118 | 126
  Week 2, Item 5 | 4.28 (1.40) | 4.63 (1.35) | 4.43 (1.29)
  Week 2, Item 6: number analyzed (Participants) | 145 | 118 | 126
  Week 2, Item 6 | 3.79 (1.31) | 4.19 (1.46) | 4.06 (1.31)
  Week 2, Item 7: number analyzed (Participants) | 145 | 118 | 126
  Week 2, Item 7 | 4.85 (1.71) | 5.31 (1.67) | 5.19 (1.64)
  Week 2, Total: number analyzed (Participants) | 145 | 118 | 126
  Week 2, Total | 29.55 (6.93) | 31.57 (7.34) | 30.94 (6.51)
  Week 3, Item 1: number analyzed (Participants) | 143 | 122 | 150
  Week 3, Item 1 | 3.94 (1.46) | 4.14 (1.60) | 4.09 (1.47)
  Week 3, Item 2: number analyzed (Participants) | 143 | 122 | 150
  Week 3, Item 2 | 3.98 (1.41) | 4.14 (1.52) | 4.25 (1.52)
  Week 3, Item 3: number analyzed (Participants) | 143 | 122 | 150
  Week 3, Item 3 | 4.20 (1.44) | 4.13 (1.50) | 4.10 (1.55)
  Week 3, Item 4: number analyzed (Participants) | 143 | 122 | 150
  Week 3, Item 4 | 5.16 (1.56) | 5.33 (1.45) | 5.51 (1.51)
  Week 3, Item 5: number analyzed (Participants) | 143 | 122 | 150
  Week 3, Item 5 | 4.44 (1.45) | 4.75 (1.45) | 4.73 (1.45)
  Week 3, Item 6: number analyzed (Participants) | 143 | 122 | 150
  Week 3, Item 6 | 3.94 (1.48) | 4.46 (1.59) | 4.51 (1.35)
  Week 3, Item 7: number analyzed (Participants) | 143 | 122 | 150
  Week 3, Item 7 | 4.80 (1.79) | 5.48 (1.65) | 5.43 (1.68)
  Week 3, Total: number analyzed (Participants) | 143 | 122 | 150
  Week 3, Total | 30.46 (7.48) | 32.43 (7.19) | 32.62 (7.20)
  Week 4, Item 1: number analyzed (Participants) | 135 | 113 | 133
  Week 4, Item 1 | 4.06 (1.51) | 4.29 (1.60) | 4.30 (1.59)
  Week 4, Item 2: number analyzed (Participants) | 135 | 113 | 133
  Week 4, Item 2 | 4.15 (1.41) | 4.40 (1.48) | 4.52 (1.52)
  Week 4, Item 3: number analyzed (Participants) | 135 | 113 | 133
  Week 4, Item 3 | 4.20 (1.62) | 4.01 (1.51) | 4.43 (1.51)
  Week 4, Item 4: number analyzed (Participants) | 135 | 113 | 133
  Week 4, Item 4 | 5.10 (1.59) | 5.32 (1.67) | 5.40 (1.59)
  Week 4, Item 5: number analyzed (Participants) | 135 | 113 | 133
  Week 4, Item 5 | 4.48 (1.48) | 4.87 (1.47) | 4.91 (1.39)
  Week 4, Item 6: number analyzed (Participants) | 135 | 113 | 133
  Week 4, Item 6 | 4.01 (1.49) | 4.58 (1.52) | 4.62 (1.50)
  Week 4, Item 7: number analyzed (Participants) | 135 | 113 | 133
  Week 4, Item 7 | 4.93 (1.70) | 5.53 (1.60) | 5.44 (1.76)
  Week 4, Total: number analyzed (Participants) | 135 | 113 | 133
  Week 4, Total | 30.93 (7.59) | 33.00 (7.67) | 33.62 (7.81)
  Week 8, Item 1: number analyzed (Participants) | 124 | 124 | 146
  Week 8, Item 1 | 4.23 (1.57) | 4.71 (1.59) | 4.60 (1.64)
  Week 8, Item 2: number analyzed (Participants) | 124 | 124 | 146
  Week 8, Item 2 | 4.44 (1.46) | 4.70 (1.50) | 4.61 (1.53)
  Week 8, Item 3: number analyzed (Participants) | 124 | 124 | 146
  Week 8, Item 3 | 4.01 (1.57) | 4.44 (1.72) | 4.36 (1.63)
  Week 8, Item 4: number analyzed (Participants) | 124 | 124 | 146
  Week 8, Item 4 | 5.37 (1.53) | 5.59 (1.41) | 5.40 (1.66)
  Week 8, Item 5: number analyzed (Participants) | 124 | 124 | 146
  Week 8, Item 5 | 4.75 (1.46) | 5.10 (1.44) | 4.95 (1.44)
  Week 8, Item 6: number analyzed (Participants) | 124 | 124 | 146
  Week 8, Item 6 | 4.42 (1.51) | 4.83 (1.57) | 4.72 (1.54)
  Week 8, Item 7: number analyzed (Participants) | 124 | 124 | 146
  Week 8, Item 7 | 5.28 (1.68) | 5.73 (1.57) | 5.60 (1.63)
  Week 8, Total: number analyzed (Participants) | 124 | 124 | 146
  Week 8, Total | 32.49 (8.00) | 35.09 (7.72) | 34.24 (8.24)
Statistical Analysis 1: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference in total score at week 1; Test type: Superiority; Mean Difference (Final Values) = 0.96
Statistical Analysis 2: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference in total score at week 2; Test type: Superiority; Mean Difference (Final Values) = 0.63
Statistical Analysis 3: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference in total score at week 3; Test type: Superiority; Mean Difference (Final Values) = 0.19
Statistical Analysis 4: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference in total score at week 4; Test type: Superiority; Mean Difference (Final Values) = 0.62
Statistical Analysis 5: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference in total score at week 8; Test type: Superiority; Mean Difference (Final Values) = 0.85
Statistical Analysis 6: Comparison: Study 2, Control vs Study 2, DIY Tool With AI; Mean difference in total score at week 1; Test type: Superiority; Mean Difference (Final Values) = 0.41
Statistical Analysis 7: Comparison: Study 2, Control vs Study 2, DIY Tool With AI; Mean difference in total score at week 2; Test type: Superiority; Mean Difference (Final Values) = 1.39
Statistical Analysis 8: Comparison: Study 2, Control vs Study 2, DIY Tool With AI; Mean difference in total score at week 3; Test type: Superiority; Mean Difference (Final Values) = 2.16
Statistical Analysis 9: Comparison: Study 2, Control vs Study 2, DIY Tool With AI; Mean difference in total score at week 4; Test type: Superiority; Mean Difference (Final Values) = 2.69
Statistical Analysis 10: Comparison: Study 2, Control vs Study 2, DIY Tool With AI; Mean difference in total score at week 8; Test type: Superiority; Mean Difference (Final Values) = 1.75

9. Primary Outcome: Study 2: Tool Mechanisms
Description: Tool Mechanisms is measured using 4 items about reframing. The items measure relatability/believability, helpfulness, memorability, and learnability on a scale of 1 (strongly disagree) to 5 (strongly agree). Total scores range from 4 to 20, with higher scores indicating better outcomes after using a Do-It-Yourself (DIY) tool. Scores will be assessed using mean item-level and total scores.
  Item 1: I believe in the reframe I came up with; Item 2: The reframe helped me deal with the thought I was struggling with; Item 3: I will remember this reframe the next time I experience this thought; Item 4: By doing this activity, I learned how I can deal with future negative thoughts
Time Frame: Week 1, Week 2, Week 3, Week 4
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study 2, DIY Tool Without AI | Study 2, DIY Tool With AI
Number analyzed (Participants) | 224 | 249
units on a scale
  Week 1, Item 1: number analyzed (Participants) | 215 | 236
  Week 1, Item 1 | 4.15 (0.99) | 4.06 (1.01)
  Week 1, Item 2: number analyzed (Participants) | 215 | 236
  Week 1, Item 2 | 3.93 (1.09) | 3.95 (1.10)
  Week 1, Item 3: number analyzed (Participants) | 215 | 236
  Week 1, Item 3 | 3.59 (1.21) | 3.68 (1.17)
  Week 1, Item 4: number analyzed (Participants) | 215 | 236
  Week 1, Item 4 | 3.85 (1.12) | 3.88 (1.15)
  Week 1, Total: number analyzed (Participants) | 215 | 236
  Week 1, Total | 15.51 (3.45) | 15.58 (3.63)
  Week 2, Item 1: number analyzed (Participants) | 157 | 179
  Week 2, Item 1 | 4.07 (1.05) | 4.11 (1.00)
  Week 2, Item 2: number analyzed (Participants) | 157 | 179
  Week 2, Item 2 | 3.91 (1.09) | 4.04 (1.02)
  Week 2, Item 3: number analyzed (Participants) | 157 | 179
  Week 2, Item 3 | 3.73 (1.18) | 3.89 (1.09)
  Week 2, Item 4: number analyzed (Participants) | 157 | 179
  Week 2, Item 4 | 3.86 (1.14) | 3.95 (1.08)
  Week 2, Total: number analyzed (Participants) | 157 | 179
  Week 2, Total | 15.57 (3.61) | 15.99 (3.47)
  Week 3, Item 1: number analyzed (Participants) | 145 | 176
  Week 3, Item 1 | 4.28 (0.92) | 4.05 (1.04)
  Week 3, Item 2: number analyzed (Participants) | 145 | 176
  Week 3, Item 2 | 4.10 (0.99) | 4.01 (1.08)
  Week 3, Item 3: number analyzed (Participants) | 145 | 176
  Week 3, Item 3 | 3.84 (1.17) | 3.82 (1.21)
  Week 3, Item 4: number analyzed (Participants) | 145 | 176
  Week 3, Item 4 | 4.01 (1.10) | 3.95 (1.12)
  Week 3, Total: number analyzed (Participants) | 145 | 176
  Week 3, Total | 16.23 (3.43) | 15.83 (3.79)
  Week 4, Item 1: number analyzed (Participants) | 125 | 157
  Week 4, Item 1 | 4.23 (0.95) | 3.98 (1.08)
  Week 4, Item 2: number analyzed (Participants) | 125 | 157
  Week 4, Item 2 | 4.07 (1.01) | 3.95 (1.11)
  Week 4, Item 3: number analyzed (Participants) | 125 | 157
  Week 4, Item 3 | 3.81 (1.19) | 3.84 (1.16)
  Week 4, Item 4: number analyzed (Participants) | 125 | 157
  Week 4, Item 4 | 3.92 (1.17) | 3.93 (1.11)
  Week 4, Total: number analyzed (Participants) | 125 | 157
  Week 4, Total | 16.03 (3.53) | 15.71 (3.90)
Statistical Analysis 1: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference in total score at week 1; Test type: Superiority; Mean Difference (Final Values) = 0.07
Statistical Analysis 2: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference in total score at week 2; Test type: Superiority; Mean Difference (Final Values) = 0.42
Statistical Analysis 3: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference in total score at week 3; Test type: Superiority; Mean Difference (Final Values) = 0.40
Statistical Analysis 4: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference in total score at week 4; Test type: Superiority; Mean Difference (Final Values) = 0.32

10. Primary Outcome: Study 2: Tool Mechanisms (Part 2)
Description: Tool Mechanisms (Part 2) is measured using 2 items about belief change and emotion change on a scale of -7 to 7. Total scores range from -14 to 14, with higher scores indicating stronger beliefs and emotions after completing a DIY tool. Note: this also includes 1 qualitative question; not included here. Scores will be assessed using mean item-level and total scores.
  Item 1: After doing this activity, how strongly do you believe in your original thought? Item 2: After doing this activity, how strong is your emotion?
Time Frame: Week 1, Week 2, Week 3, Week 4
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study 2, DIY Tool Without AI | Study 2, DIY Tool With AI
Number analyzed (Participants) | 224 | 249
units on a scale
  Week 1, Item 1: number analyzed (Participants) | 215 | 236
  Week 1, Item 1 | 1.38 (1.50) | 1.42 (1.58)
  Week 1, Item 2: number analyzed (Participants) | 215 | 236
  Week 1, Item 2 | 1.65 (1.47) | 1.62 (1.50)
  Week 1, Total: number analyzed (Participants) | 215 | 236
  Week 1, Total | 3.03 (2.69) | 3.04 (2.79)
  Week 2, Item 1: number analyzed (Participants) | 157 | 179
  Week 2, Item 1 | 1.27 (1.47) | 1.46 (1.47)
  Week 2, Item 2: number analyzed (Participants) | 157 | 179
  Week 2, Item 2 | 1.44 (1.55) | 1.61 (1.44)
  Week 2, Total: number analyzed (Participants) | 157 | 179
  Week 2, Total | 2.71 (2.79) | 3.08 (2.66)
  Week 3, Item 1: number analyzed (Participants) | 145 | 176
  Week 3, Item 1 | 1.36 (1.62) | 1.40 (1.47)
  Week 3, Item 2: number analyzed (Participants) | 145 | 176
  Week 3, Item 2 | 1.56 (1.74) | 1.50 (1.59)
  Week 3, Total: number analyzed (Participants) | 145 | 176
  Week 3, Total | 2.91 (3.09) | 2.90 (2.84)
  Week 4, Item 1: number analyzed (Participants) | 125 | 157
  Week 4, Item 1 | 1.51 (1.65) | 1.51 (1.60)
  Week 4, Item 2: number analyzed (Participants) | 125 | 157
  Week 4, Item 2 | 1.76 (1.75) | 1.47 (1.51)
  Week 4, Total: number analyzed (Participants) | 125 | 157
  Week 4, Total | 3.27 (3.13) | 2.98 (2.90)
Statistical Analysis 1: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference in total score at week 1; Test type: Superiority; Mean Difference (Final Values) = 0.01
Statistical Analysis 2: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference in total score at week 2; Test type: Superiority; Mean Difference (Final Values) = 0.37
Statistical Analysis 3: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference in total score at week 3; Test type: Superiority; Mean Difference (Final Values) = 0.01
Statistical Analysis 4: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference in total score at week 4; Test type: Superiority; Mean Difference (Final Values) = 0.29

11. Primary Outcome: Study 2: DIY Skill Use: Competencies of Cognitive Therapy Scale - Self-Report
Description: The Competencies of Cognitive Therapy Scale will be used to ask participants about how much they have used specific strategies to cope with negative moods, primarily negative automatic thoughts, in the last 4 weeks. The current study will use items 20, 28, 21, 6, 24, and 11. Items are rated from 1 (not at all) to 7 (completely). Total scores range from 6 to 42. Higher scores indicate better outcomes. Scores will be assessed using mean item-level and total scores. Note: also includes 3 qualitative questions; not included here. Themes:
  Item 20: re-evaluating the situation; Item 28: taking time to step back and considering that negative thoughts might be inaccurate; Item 21: actively working to develop more rational views; Item 6: having a specific action plan of things they could do to cope; Item 24: taking time to consider other factors that may have been involved; Item 11: taking note of what they were thinking and working to develop a more balanced view
Time Frame: Week 1, Week 2, Week 3, Week 4, Week 8
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study 2, Control | Study 2, DIY Tool Without AI | Study 2, DIY Tool With AI
Number analyzed (Participants) | 210 | 188 | 212
units on a scale
  Week 1, Item 20: number analyzed (Participants) | 187 | 163 | 177
  Week 1, Item 20 | 3.43 (1.52) | 3.77 (1.50) | 3.68 (1.49)
  Week 1, Item 28: number analyzed (Participants) | 187 | 164 | 177
  Week 1, Item 28 | 3.56 (1.62) | 3.85 (1.55) | 3.86 (1.59)
  Week 1, Item 21: number analyzed (Participants) | 187 | 164 | 177
  Week 1, Item 21 | 3.56 (1.64) | 3.95 (1.56) | 3.80 (1.63)
  Week 1, Item 6: number analyzed (Participants) | 187 | 164 | 177
  Week 1, Item 6 | 2.82 (1.58) | 3.51 (1.70) | 3.26 (1.56)
  Week 1, Item 24: number analyzed (Participants) | 187 | 164 | 177
  Week 1, Item 24 | 3.38 (1.71) | 3.79 (1.71) | 3.84 (1.63)
  Week 1, Item 11: number analyzed (Participants) | 187 | 164 | 177
  Week 1, Item 11 | 3.29 (1.62) | 3.76 (1.55) | 3.58 (1.58)
  Week 1, Total: number analyzed (Participants) | 187 | 163 | 177
  Week 1, Total | 20.04 (7.79) | 22.60 (7.61) | 22.02 (7.95)
  Week 2, Item 20: number analyzed (Participants) | 145 | 118 | 124
  Week 2, Item 20 | 3.94 (1.52) | 4.00 (1.56) | 4.05 (1.55)
  Week 2, Item 28: number analyzed (Participants) | 144 | 118 | 124
  Week 2, Item 28 | 3.94 (1.60) | 4.06 (1.57) | 4.10 (1.55)
  Week 2, Item 21: number analyzed (Participants) | 145 | 118 | 124
  Week 2, Item 21 | 3.90 (1.68) | 4.13 (1.55) | 3.98 (1.63)
  Week 2, Item 6: number analyzed (Participants) | 145 | 118 | 124
  Week 2, Item 6 | 3.39 (1.56) | 3.84 (1.72) | 3.80 (1.59)
  Week 2, Item 24: number analyzed (Participants) | 145 | 118 | 124
  Week 2, Item 24 | 3.74 (1.63) | 4.07 (1.60) | 3.99 (1.60)
  Week 2, Item 11: number analyzed (Participants) | 145 | 118 | 124
  Week 2, Item 11 | 3.70 (1.63) | 3.77 (1.61) | 3.86 (1.64)
  Week 2, Total: number analyzed (Participants) | 144 | 118 | 124
  Week 2, Total | 22.60 (7.91) | 23.86 (7.90) | 23.78 (8.30)
  Week 3, Item 20: number analyzed (Participants) | 143 | 121 | 150
  Week 3, Item 20 | 3.87 (1.70) | 4.22 (1.60) | 4.31 (1.66)
  Week 3, Item 28: number analyzed (Participants) | 143 | 121 | 150
  Week 3, Item 28 | 3.87 (1.66) | 4.26 (1.73) | 4.47 (1.56)
  Week 3, Item 21: number analyzed (Participants) | 143 | 121 | 150
  Week 3, Item 21 | 3.69 (1.61) | 4.04 (1.65) | 4.33 (1.69)
  Week 3, Item 6: number analyzed (Participants) | 143 | 121 | 150
  Week 3, Item 6 | 3.41 (1.76) | 3.91 (1.68) | 4.17 (1.72)
  Week 3, Item 24: number analyzed (Participants) | 143 | 121 | 150
  Week 3, Item 24 | 3.82 (1.76) | 4.21 (1.77) | 4.37 (1.68)
  Week 3, Item 11: number analyzed (Participants) | 143 | 121 | 150
  Week 3, Item 11 | 3.71 (1.76) | 4.15 (1.68) | 4.38 (1.63)
  Week 3, Total: number analyzed (Participants) | 143 | 121 | 150
  Week 3, Total | 22.36 (8.67) | 24.79 (8.62) | 26.03 (8.63)
  Week 4, Item 20: number analyzed (Participants) | 132 | 113 | 133
  Week 4, Item 20 | 3.69 (1.72) | 4.26 (1.78) | 4.39 (1.77)
  Week 4, Item 28: number analyzed (Participants) | 131 | 113 | 133
  Week 4, Item 28 | 3.71 (1.82) | 4.24 (1.78) | 4.34 (1.75)
  Week 4, Item 21: number analyzed (Participants) | 132 | 113 | 133
  Week 4, Item 21 | 3.42 (1.72) | 4.30 (1.72) | 4.20 (1.72)
  Week 4, Item 6: number analyzed (Participants) | 132 | 113 | 133
  Week 4, Item 6 | 3.36 (1.89) | 3.92 (1.89) | 4.06 (1.81)
  Week 4, Item 24: number analyzed (Participants) | 132 | 113 | 133
  Week 4, Item 24 | 3.61 (1.86) | 4.32 (1.94) | 4.33 (1.88)
  Week 4, Item 11: number analyzed (Participants) | 132 | 113 | 133
  Week 4, Item 11 | 3.61 (1.82) | 4.18 (1.91) | 4.36 (1.86)
  Week 4, Total: number analyzed (Participants) | 131 | 113 | 133
  Week 4, Total | 21.46 (9.33) | 25.21 (9.66) | 25.68 (9.63)
  Week 8, Item 20: number analyzed (Participants) | 123 | 123 | 145
  Week 8, Item 20 | 3.90 (1.91) | 4.24 (1.89) | 4.34 (1.89)
  Week 8, Item 28: number analyzed (Participants) | 123 | 123 | 145
  Week 8, Item 28 | 4.02 (1.94) | 4.55 (1.84) | 4.66 (1.84)
  Week 8, Item 21: number analyzed (Participants) | 123 | 123 | 145
  Week 8, Item 21 | 3.93 (1.86) | 4.28 (2.00) | 4.32 (1.88)
  Week 8, Item 6: number analyzed (Participants) | 123 | 123 | 145
  Week 8, Item 6 | 3.98 (1.87) | 4.33 (1.90) | 4.23 (1.92)
  Week 8, Item 24: number analyzed (Participants) | 123 | 123 | 145
  Week 8, Item 24 | 4.36 (2.00) | 4.51 (1.94) | 4.54 (1.93)
  Week 8, Item 11: number analyzed (Participants) | 123 | 123 | 145
  Week 8, Item 11 | 4.23 (1.85) | 4.54 (1.91) | 4.41 (2.01)
  Week 8, Total: number analyzed (Participants) | 123 | 123 | 145
  Week 8, Total | 24.42 (9.80) | 26.46 (10.12) | 26.49 (10.31)
Statistical Analysis 1: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference in total score at week 1; Test type: Superiority; Mean Difference (Final Values) = 0.58
Statistical Analysis 2: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference in total score at week 2; Test type: Superiority; Mean Difference (Final Values) = 0.08
Statistical Analysis 3: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference in total score at week 3; Test type: Superiority; Mean Difference (Final Values) = 1.24
Statistical Analysis 4: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference in total score at week 4; Test type: Superiority; Mean Difference (Final Values) = 0.47
Statistical Analysis 5: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference in total score at week 8; Test type: Superiority; Mean Difference (Final Values) = 0.03
Statistical Analysis 6: Comparison: Study 2, Control vs Study 2, DIY Tool With AI; Mean difference in total score at week 1; Test type: Superiority; Mean Difference (Final Values) = 1.98
Statistical Analysis 7: Comparison: Study 2, Control vs Study 2, DIY Tool With AI; Mean difference in total score at week 2; Test type: Superiority; Mean Difference (Final Values) = 1.18
Statistical Analysis 8: Comparison: Study 2, Control vs Study 2, DIY Tool With AI; Mean difference in total score at week 3; Test type: Superiority; Mean Difference (Final Values) = 3.67
Statistical Analysis 9: Comparison: Study 2, Control vs Study 2, DIY Tool With AI; Mean difference in total score at week 4; Test type: Superiority; Mean Difference (Final Values) = 4.22
Statistical Analysis 10: Comparison: Study 2, Control vs Study 2, DIY Tool With AI; Mean difference in total score at week 8; Test type: Superiority; Mean Difference (Final Values) = 2.07

12. Primary Outcome: Long-term Adoption of the Intervention
Description: We measure long-term adoption of the Intervention using an 8-item scale assessing attitudes and behaviors related to engaging with and adopting a mental health intervention focused on reframing negative thoughts. Each item is scored on a scale from 1 to 10. Higher scores indicate greater comfort, likelihood, willingness, excitement, or impact, depending on the item. Specifically, the items assess comfort with attending therapy (Item 1), working with a therapist on reframing (Item 2), and discussing negative thoughts (Item 3); likelihood of seeking mental health information (Item 4); willingness to commit to practicing reframing (Item 5); excitement about learning a new mental health skill (Item 6); the impact of negative thoughts on life (Item 7); and likelihood of recommending the intervention to a friend (Item 8). Scores will be assessed using mean item-level scores. No statistical analysis conducted.
Time Frame: Week 5
Population: Participants who completed week 5.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study 2, Control | Study 2, DIY Tool Without AI | Study 2, DIY Tool With AI
Number analyzed (Participants) | 166 | 137 | 155
units on a scale
  Item 1 | 7.04 (2.65) | 6.82 (2.94) | 6.94 (2.77)
  Item 2 | 7.39 (2.38) | 7.17 (2.59) | 7.28 (2.63)
  Item 3 | 5.55 (2.76) | 5.62 (2.85) | 5.45 (2.73)
  Item 4 | 8.15 (2.13) | 8.28 (2.16) | 8.07 (2.38)
  Item 5 | 7.63 (2.10) | 7.92 (2.02) | 7.78 (2.31)
  Item 6 | 7.51 (2.37) | 7.99 (2.32) | 7.65 (2.32)
  Item 7 | 7.73 (1.78) | 7.62 (1.87) | 7.63 (1.84)
  Item 8 | 5.54 (2.83) | 6.05 (2.93) | 5.55 (2.82)

13. Primary Outcome: Hopefulness
Description: Hopefulness is measured using a single item (How hopeful do you feel about the future?). Scores will be assessed using mean item-level scores. Scores range from 1 to 7, with higher scores indicating better outcomes (more hopefulness). No statistical analysis (this item was merged with emotion mechanisms).
Time Frame: Week 1, Week 2, Week 3, Week 4, Week 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study 2, Control | Study 2, DIY Tool Without AI | Study 2, DIY Tool With AI
Number analyzed (Participants) | 219 | 196 | 219
units on a scale
  Week 1: number analyzed (Participants) | 195 | 172 | 182
  Week 1 | 3.66 (1.28) | 3.87 (1.43) | 3.77 (1.23)
  Week 2: number analyzed (Participants) | 145 | 118 | 126
  Week 2 | 3.73 (1.37) | 4.03 (1.53) | 3.84 (1.36)
  Week 3: number analyzed (Participants) | 143 | 122 | 150
  Week 3 | 3.94 (1.46) | 4.14 (1.60) | 4.09 (1.47)
  Week 4: number analyzed (Participants) | 135 | 113 | 133
  Week 4 | 4.06 (1.51) | 4.29 (1.60) | 4.30 (1.59)
  Week 8: number analyzed (Participants) | 124 | 124 | 146
  Week 8 | 4.23 (1.57) | 4.71 (1.59) | 4.60 (1.64)

14. Secondary Outcome: Study 2: Patient Health Questionnaire-9 (PHQ-9)
Description: The Patient Health Questionnaire-9 (PHQ-9) consists of 9 depression items. Each item is associated with a Diagnostic and Statistical Manual (DSM) symptom of depression. Participants rate whether or not they have experienced the symptom over the last two weeks, with severity ratings of 0 to 3. Total scores range from 0 to 27, with higher scores indicating greater severity of depression symptoms. It is one of the few measures that is brief (it takes less than one minute to give) and has been found to have excellent sensitivity to change over time.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study 2, Control | Study 2, DIY Tool Without AI | Study 2, DIY Tool With AI
Number analyzed (Participants) | 269 | 272 | 298
units on a scale
  Baseline | 17.69 (4.66) | 17.66 (4.86) | 17.97 (4.68)
  Week 1: number analyzed (Participants) | 197 | 172 | 183
  Week 1 | 14.50 (5.03) | 14.88 (5.83) | 15.17 (5.26)
  Week 2: number analyzed (Participants) | 148 | 118 | 127
  Week 2 | 13.58 (5.52) | 12.92 (5.81) | 12.80 (5.20)
  Week 3: number analyzed (Participants) | 146 | 123 | 151
  Week 3 | 12.84 (6.22) | 12.79 (6.14) | 12.66 (5.97)
  Week 4: number analyzed (Participants) | 138 | 115 | 135
  Week 4 | 11.51 (6.06) | 12.72 (6.79) | 11.04 (6.21)
  Week 8: number analyzed (Participants) | 130 | 127 | 146
  Week 8 | 10.58 (6.66) | 10.66 (6.50) | 10.82 (6.88)
Statistical Analysis 1: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference at baseline; Test type: Superiority; Mean Difference (Final Values) = 0.31
Statistical Analysis 2: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference at week 1; Test type: Superiority; Mean Difference (Final Values) = 0.29
Statistical Analysis 3: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference at week 2; Test type: Superiority; Mean Difference (Final Values) = 0.12
Statistical Analysis 4: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference at week 3; Test type: Superiority; Mean Difference (Final Values) = 0.13
Statistical Analysis 5: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference at week 4; Test type: Superiority; Mean Difference (Final Values) = 1.68
Statistical Analysis 6: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference at week 8; Test type: Superiority; Mean Difference (Final Values) = 0.16
Statistical Analysis 7: Comparison: Study 2, Control vs Study 2, DIY Tool With AI; Mean difference at baseline; Test type: Superiority; Mean Difference (Final Values) = 0.28
Statistical Analysis 8: Comparison: Study 2, Control vs Study 2, DIY Tool With AI; Mean difference at week 1; Test type: Superiority; Mean Difference (Final Values) = 0.67
Statistical Analysis 9: Comparison: Study 2, Control vs Study 2, DIY Tool With AI; Mean difference at week 2; Test type: Superiority; Mean Difference (Final Values) = 0.78
Statistical Analysis 10: Comparison: Study 2, Control vs Study 2, DIY Tool With AI; Mean difference at week 3; Test type: Superiority; Mean Difference (Final Values) = 0.18
Statistical Analysis 11: Comparison: Study 2, Control vs Study 2, DIY Tool With AI; Mean difference at week 4; Test type: Superiority; Mean Difference (Final Values) = 0.47
Statistical Analysis 12: Comparison: Study 2, Control vs Study 2, DIY Tool With AI; Mean difference at week 8; Test type: Superiority; Mean Difference (Final Values) = 0.24

15. Secondary Outcome: Study 2: Generalized Anxiety Disorder-7 (GAD-7)
Description: The Generalized Anxiety Disorder-7 (GAD-7) is a 7- item screener for generalized anxiety. It consists of items related to Generalized Anxiety Disorder (GAD). Participants rate how much anxiety they have experienced in the last two weeks on a scale of 0 to 3. Total scores range from 0 to 21, with higher scores indicating greater severity of anxiety symptoms. The scale is a valid screener for GAD.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Study 2, Control | Study 2, DIY Tool Without AI | Study 2, DIY Tool With AI
Number analyzed (Participants) | 268 | 272 | 298
units on a scale
  Baseline: number analyzed (Participants) | 268 | 271 | 298
  Baseline | 14.29 (4.62) | 14.56 (4.14) | 14.38 (4.65)
  Week 1: number analyzed (Participants) | 196 | 171 | 183
  Week 1 | 12.43 (4.71) | 12.84 (4.93) | 12.69 (5.36)
  Week 2: number analyzed (Participants) | 145 | 118 | 126
  Week 2 | 11.28 (4.81) | 11.46 (5.58) | 11.23 (5.23)
  Week 3: number analyzed (Participants) | 143 | 122 | 150
  Week 3 | 10.83 (5.57) | 11.51 (5.79) | 11.13 (5.61)
  Week 4: number analyzed (Participants) | 135 | 113 | 133
  Week 4 | 10.10 (5.74) | 11.06 (6.08) | 9.80 (5.64)
  Week 8: number analyzed (Participants) | 124 | 124 | 146
  Week 8 | 9.22 (5.72) | 9.36 (6.15) | 9.62 (6.35)
Statistical Analysis 1: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference at baseline; Test type: Superiority; Mean Difference (Final Values) = 0.18
Statistical Analysis 2: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference at week 1; Test type: Superiority; Mean Difference (Final Values) = 0.15
Statistical Analysis 3: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference at week 2; Test type: Superiority; Mean Difference (Final Values) = 0.23
Statistical Analysis 4: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference at week 3; Test type: Superiority; Mean Difference (Final Values) = 0.38
Statistical Analysis 5: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference at week 4; Test type: Superiority; Mean Difference (Final Values) = 1.26
Statistical Analysis 6: Comparison: Study 2, DIY Tool Without AI vs Study 2, DIY Tool With AI; Mean difference at week 8; Test type: Superiority; Mean Difference (Final Values) = 0.26
Statistical Analysis 7: Comparison: Study 2, Control vs Study 2, DIY Tool With AI; Mean difference at baseline; Test type: Superiority; Mean Difference (Final Values) = 0.09
Statistical Analysis 8: Comparison: Study 2, Control vs Study 2, DIY Tool With AI; Mean difference at week 1; Test type: Superiority; Mean Difference (Final Values) = 0.26
Statistical Analysis 9: Comparison: Study 2, Control vs Study 2, DIY Tool With AI; Mean difference at week 2; Test type: Superiority; Mean Difference (Final Values) = 0.05
Statistical Analysis 10: Comparison: Study 2, Control vs Study 2, DIY Tool With AI; Mean difference at week 3; Test type: Superiority; Mean Difference (Final Values) = 0.30
Statistical Analysis 11: Comparison: Study 2, Control vs Study 2, DIY Tool With AI; Mean difference at week 4; Test type: Superiority; Mean Difference (Final Values) = 0.30
Statistical Analysis 12: Comparison: Study 2, Control vs Study 2, DIY Tool With AI; Mean difference at week 8; Test type: Superiority; Mean Difference (Final Values) = 0.40

ADVERSE EVENTS:
Time Frame: Study 1: Adverse events were collected for the entirety of time users spent in a single session while using the Mental Health America (MHA) website, from the time that they entered the MHA website to the time that they exited the website, or when their session ended. Adverse events were collected throughout the entirety of the study's 3-month duration. Study 2: Adverse events were collected for the entirety of time patients were in the study from baseline to 8 week follow-up.
Arm/Group | Study 1, Demographic Survey | Study 1, Next Steps Survey | Study 1, Demographic Survey + Generic Response + Generic Resources | Study 1, Demographic Survey + Generic Response + Tailored Resources by Demographics | Study 1, Next Steps Survey + Generic Response + Generic Resources | Study 1, Next Steps Survey + Generic Response + Tailored Resources by Desired Resources | Study 1, Next Steps Survey + Tailored Response + Generic Resources | Study 1, Next Steps Survey + Tailored Response + Tailored Resources by Desired Resources | Study 2, Control | Study 2, DIY Tool Without AI | Study 2, DIY Tool With AI
All-Cause Mortality (participants affected / at risk) | 0/2490 | 0/2367 | 0/19250 | 0/19240 | 0/8743 | 0/8636 | 0/8454 | 0/8371 | 0/269 | 0/272 | 0/298
Serious Adverse Events (participants affected / at risk) | 0/2490 | 0/2367 | 0/19250 | 0/19240 | 0/8743 | 0/8636 | 0/8454 | 0/8371 | 0/269 | 0/272 | 0/298
Other Adverse Events (participants affected / at risk) | 0/2490 | 0/2367 | 0/19250 | 0/19240 | 0/8743 | 0/8636 | 0/8454 | 0/8371 | 0/269 | 0/272 | 0/298

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-07-03): https://cdn.clinicaltrials.gov/large-docs/60/NCT04507360/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-03): https://cdn.clinicaltrials.gov/large-docs/60/NCT04507360/SAP_001.pdf
  • Informed Consent Form (2023-11-14): https://cdn.clinicaltrials.gov/large-docs/60/NCT04507360/ICF_002.pdf